CLINICAL TRIAL: NCT00647244
Title: Efficacy and Safety of Switching From AZT to Tenofovir
Brief Title: Efficacy and Safety of Switching From Retrovir to Tenofovir or Abacavir in HIV-infected Patients
Acronym: SWAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Alex Lund Laursen, MD, PhD, DmSC, Department of Infectious Diseases, Aarhus University Hospital, Denmark
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKS-HIV-002; EudraCT2007-004372-39
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-12

CONDITIONS: HIV Infections
Keywords: Tenofovir; Abacavir; Antiretroviral therapy; HIV; Nucleoside analogue reverse transcriptase inhibitor
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Tenofovir
  Interventions: Drug: Tenofovir disoproxil fumarate
- 2 (Active Comparator): Abacavir
  Interventions: Drug: Abacavir

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate — Tenofovir disoproxil 245 mg oral tablet once daily
  Arms: 1
Drug: Abacavir — Abacavir 300 mg oral tablet twice daily
  Arms: 2

SUMMARY:
To evaluate the efficacy and safety of switching from Retrovir to Tenofovir or Abacavir in HIV-infected patients

ELIGIBILITY:
Inclusion Criteria:

* HIV-infection with undetectable viral load
* Antiretroviral treatment including Retrovir for more than three months
* If fertile female: Negative pregnancy test and use of safe contraception
* Negative HBs-antigen titer

Exclusion Criteria:

* Prior treatment with abacavir or tenofovir
* Resistance towards abacavir or tenofovir
* Tissue type HLA-B5701
* Renal disease
* Diabetes Mellitus
* Osteoporosis
* Pregnant or lactating subjects
* Intravenous drug abuse
* Hypersensitivity towards drugs or active ingredient used
* ALAT > 5 times upper normal level
* Current alcohol or substance abuse judged by the Investigator to potentially interfere with subject compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Renal function measured by Cystatin-C and creatinine clearance | Weeks 0, 4, 8, 12, 24, 24, 48, 96
Levels of renal tubule function markers in blood and urine | Weeks 0, 12, 24, 48, 96
Bone mass assessed by DEXA | Weeks 0, 24, 48, 96
Levels of bone turnover markers in blood and urine | Weeks 0, 12, 24, 48, 96
Insulin resistance | Weeks 0, 12, 24, 48, 96
Changes in body composition assessed by patient questionnaire and standardized examination by physician | Weeks 0, 12, 24, 48, 96
Changes in subcutaneous adipose tissue assessed by DEXA | Week 0, 24, 48, 96

SECONDARY OUTCOMES:
Patients with viral load < 40 copies/ml | Weeks 0, 4, 8, 12, 24, 48, 96
CD-4 cell count | Weeks 0, 4, 8, 12, 24, 48, 96
Fasting triglycerides, HDL and LDL | Weeks 0, 12, 24, 48, 96
Development of resistance mutations | Weeks 0, 12, 24, 48, 96
Development of adverse events and serious adverse events | Weeks 0, 4, 8, 12, 24, 48, 96

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Århus N, Denmark

REFERENCES:
- [Derived] Rasmussen TA, Jensen D, Tolstrup M, Nielsen US, Erlandsen EJ, Birn H, Ostergaard L, Langdahl BL, Laursen AL. Comparison of bone and renal effects in HIV-infected adults switching to abacavir or tenofovir based therapy in a randomized trial. PLoS One. 2012;7(3):e32445. doi: 10.1371/journal.pone.0032445. Epub 2012 Mar 29. PMID 22479327
- [Derived] Rasmussen TA, Tolstrup M, Melchjorsen J, Frederiksen CA, Nielsen US, Langdahl BL, Ostergaard L, Laursen AL. Evaluation of cardiovascular biomarkers in HIV-infected patients switching to abacavir or tenofovir based therapy. BMC Infect Dis. 2011 Oct 4;11:267. doi: 10.1186/1471-2334-11-267. PMID 21970555